CLINICAL TRIAL: NCT01030276
Title: Placebo-controlled, Double Blind RCT on the Efficacy of Bright Light Therapy in SAD
Brief Title: Bright Light Therapy in Seasonal Affective Disorder (SAD)
Acronym: VAHAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other); ODL Terveys Oy (Unknown); Valkee Oy (Industry); University of Eastern Finland (Other)
Responsible Party: Osmo Tervonen, professor of Radiology, Institute of Diagnostics (Radiology), University of Oulu, Box 5000, FIN-90014 University of Oulu, Finland
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FI (FWA00000190) 11/2008
Record Dates: First submitted 2009-12-10; First posted 2009-12-11 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-12

CONDITIONS: Seasonal Affective Disorder
MeSH Terms: conditions — Seasonal Affective Disorder | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bright light (Experimental)
  Interventions: Other: Bright light therapy
- Inactive "placebo-light" (Placebo Comparator)
  Interventions: Other: Inactive "placebo-light"

INTERVENTIONS:
Other: Bright light therapy — Bright light therapy
  Arms: Bright light
Other: Inactive "placebo-light" — In this arm, patients will not get any bright-light therapy in a double-blind setting
  Arms: Inactive "placebo-light"

SUMMARY:
The aim of this study is to investigate the efficacy of bright light therapy in SAD. This is a placebo-controlled, double-blind randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* a patient has, according to the DSM-IV-TR, a Major depression, recurrent episode, seasonal pattern, "moderate" or "severe" (classification code 296.32 and 296.33)
* HAMD-21 (included in the SIGH-SAD) sum score is ≥ 22
* patient is over 18 years
* patient can read and understand the subject information sheet
* patient has signed the informed consent form
* patient is not pregnant

Exclusion Criteria:

* patient has a lifetime psychotic disorder
* patient has a DSM-IV Axis I disorder other than some anxiety disorder evaluated by MINI
* patient has some DSM-IV-TR Axis II disorder, which is likely to interfere with the study treatment according to the investigator
* patient has alcohol or some other substance use dependence or misuse
* life-time suicide attempt, or any thought of suicide during the last month
* patients has some unstable somatic disorder
* patient uses some medication on regular basis
* patient uses some herbal psychotropic agencies
* patient is, in the opinion of the investigator, unsuitable for any reason
* patient is a member of the site personnel or their immediate families
* patient has had bright light therapy during the current episode
* patient has some eye disease (patient can, however, be myopic or hyperopic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-03 (Estimated); Study Completion 2011-04 (Estimated)

PRIMARY OUTCOMES:
Remission as defined by the SIGH-SAD | 28 (visit window from 26 to 30 days) days after the inclusion day

SECONDARY OUTCOMES:
Decrease of the severity of symptoms as assessed by SIGH-SAD, Hamilton anxiety scale, and Beck depression inventory-21 | 28 (visit window from 26 to 30 days) days

CONTACTS AND LOCATIONS:
Locations (1):
- Research unit, ODL Terveys Oy, Albertinkatu 18 A, Oulu, Finland